CLINICAL TRIAL: NCT00389519
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel-Arm Study Assessing the Efficacy, Safety, and Dose-Response of Ramipril for the Treatment of Hypertension in Children and Adolescents
Brief Title: A Study of the Effectiveness and Safety of Ramipril in the Treatment of Hypertension in Children and Adolescents
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: A planned interim analysis was performed after approx. 240 subjects completed the trial. The study was stopped, as permitted by protocol, after the analysis.
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K726-06-4003
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Results first posted 2010-05-19 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Hypertension
Keywords: Hypertension/*etiology; Blood Pressure; Pediatric; Adolescent; Child
MeSH Terms: conditions — Hypertension | interventions — Ramipril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Placebo (Placebo Comparator): once per day
  Interventions: Drug: placebo
- ramipril low dose (Experimental): 0.3125, 0.625, or 1.25 mg once a day, based on subject weight
  Interventions: Drug: ramipril
- ramipril mid dose (Experimental): 1.25, 2.5, or 5 mg once a day, based on subject weight
  Interventions: Drug: ramipril
- ramipril high dose (Experimental): 5, 10, or 20 mg once a day, based on subject weight
  Interventions: Drug: ramipril

INTERVENTIONS:
Drug: ramipril — once a day oral ramipril capsules given for 4 weeks
  Other Names: Altace
  Arms: ramipril high dose; ramipril low dose; ramipril mid dose
Drug: placebo — once a day oral placebo capsule for 4 weeks
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the blood pressure lowering effects of ramipril, an FDA-approved drug for the treatment of hypertension in adults, in children and adolescents aged 6 to 16 years with hypertension.

DETAILED DESCRIPTION:
Information is needed on the treatment of hypertension in children and adolescents with antihypertensive drugs like ramipril. The study will assess the safety and blood pressure effects of several doses of the antihypertensive drug ramipril in children and adolescents age 6-16 years. Approximately 450 children will be given placebo, or 1 of the 3 doses of ramipril. The treatment assigned will be done by chance, like flipping a coin. Approximately 120 study centers throughout the world will participate in the trial.

Each child will complete a 1- to 4-week Screening Period where they will stop taking their current blood pressure lowering drug(s), a 4-week Treatment Period where they will receive placebo or one of the ramipril doses, and a Follow-up visit 1 week after completion of the Treatment Period. Children diagnosed with hypertension according to the fourth report on the diagnosis, evaluation and treatment of high blood pressure in children and adolescents (U.S. report), will be included in the study if their blood pressure meets certain values.

Each child will complete a minimum of 6 and up to 9 clinic visits over the course of the study during which procedures and assessments of blood pressure and safety will be performed. In addition, a child's parents/guardians will be instructed to measure their child's blood pressure at home between clinic visits.

A planned interim analysis was performed after approximately 240 subjects completed the trial. The study was stopped, as permitted by protocol, after the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Previous, documented diagnosis of hypertension, or newly diagnosed hypertension according to the fourth report on the diagnosis, evaluation and treatment of high blood pressure in children and adolescents (United States). SiSBP greater than or equal to the 95th percentile for age, gender, and height.
2. The subject can be safely withdrawn from antihypertensive medications during the screening period, and if given placebo during the treatment period in the judgment of the Investigator.
3. The subject is male or female age 6 to 16 years (inclusive), and weighs greater than or equal to 20 kg.
4. Female subjects greater than or equal to 12 years of age, or who have had greater than or equal to 1 menstruation must: (a) have a negative serum pregnancy test at screening (i.e., subject is not pregnant), (b) not be lactating, and (c) use an acceptable method of contraception.
5. Parents/guardians are able to demonstrate their ability to (a) use a home blood pressure monitor supplied for the study to monitor their child's blood pressure, and (2) mix and administer a liquid dose of study drug if needed.

Exclusion Criteria:

1. Bilateral renal artery stenosis.
2. Uncorrected coarctation of the aorta or corrected coarctation with a right arm/right leg blood pressure gradient greater than 10 mmHg.
3. Severe hypertension.
4. Renal transplantation or other previous solid organ transplantation less than 6 months prior to entering the study.
5. Subjects with nephrotic syndrome not on stable maintenance therapy of prednisone or cyclosporine.
6. A history of cardiomyopathy, clinically significant structural heart disease, or atrioventricular conduction disturbance, sick sinus syndrome, atrial flutter, atrial fibrillation, clinically significant bradycardia or an accessory bypass tract, or clinical symptoms of congestive heart failure.
7. Clinically significant hematologic, hepatobiliary, or renal disease including a Schwartz formula GFR less than 40 mL/min/1.73 m2, and/or serum potassium (K+) greater than 5.5 mEq/L.
8. History of pancreatitis (active or inactive).
9. Known sensitivity to angiotensin converting enzyme inhibitors or a history of angioneurotic edema.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 422 (Actual)
Dates: Start 2006-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (100):
- United States (39):
  - UAMS College of Medicine/ Arkansas Children's Hospital, Little Rock, Arkansas
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - Impact Clinical Research, Beverly Hills, California
  - Neufeld Medical Group, Los Angeles, California
  - Almon Clinical Research, Inc., Orange, California
  - Pediatrics in Brevard, Cocoa Beach, Florida
  - Watson Clinic Center for Research, Inc., Lakeland, Florida
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Hawaii Pacific Health, Honolulu, Hawaii
  - Nephrology and Hypertension Consultants, Park Ridge, Illinois
  - Tinley Park Pediatric Associates, Tinley Park, Illinois
  - Kosair Children's Hospital, Louisville, Kentucky
  - Louisiana State University, Shreveport, Louisiana
  - Craig Spiegel, MD, Bridgeton, Missouri
  - Impact Clinical Trials, Las Vegas, Nevada
  - Children's Heart Center, Las Vegas, Nevada
  - Premier Clinical Research Group, Toms River, New Jersey
  - SUNY Upstate Syracuse, Department of Pediatrics, Syracuse, New York
  - Hartrich Aquino & Hrab, PC, Williamsville, New York
  - Western Wake Pediatrics, Cary, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke Pediatric Clinical Research Program, Durham, North Carolina
  - North Carolina Children's and Adults Clinical Research Foundation, Sylva, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Center for Clinical and Translational Research, Columbus, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - The University of Oklahoma, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Northwest Pediatric Kidney Specialists, LLC, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Holston Medical Group, Kingsport, Tennessee
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - South East Texas Cardiology Associates, Beaumont, Texas
  - University of Texas Medical Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Huguenot Pediatrics, Midlothian, Virginia
  - Children's Specialty Group, Norfolk, Virginia
- Argentina (6):
  - Hospital de Niños "Dr. Ricardo Gutiérrez", Buenos Aires
  - Hospital General Interzonal "Dr. José Penna", Buenos Aires
  - Hospital Interzonal Especializado Materno Infantil, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital de Niños Juan Carlos Navarro, San Juan
  - Centro Infantil del Rínon, Tucomán
- Chile (4):
  - Clínica Las Condes, Santiago
  - Hospital de Niños Roberto del Rio, Santiago
  - Hospital Luis Calvo Mackena, Santiago
  - Hospital Dr. Gustavo Fricke, Viña del Mar
- Colombia (6):
  - Fundación Bios, Barranquilla
  - Fundación Cardio Infantil - Instituto de Cardiología, Bogotá
  - Hospital de San Jose, Bogotá
  - Instituto Nacional del Riñón, Bogotá
  - Hospital Pablo Tobon Uribe, Medellín
  - Hospital Universitario San Vicente de Paul, Medellín
- India (13):
  - Gujarat Kidney Foundation, Jivraj Mehta Hospital, Ahmedabad
  - Heart Care Clinic, Ahmedabad
  - St. John's Hospital, Bangalore
  - Institute of Child Health & Hospital for Children, Chennai
  - AIl India Institute medical sciences, Delhi
  - Apollo Hospital, Delhi
  - Maulana Azad Medical College and Lok Nayak Hospital, Delhi
  - Apollo Hospital Hyderabad, Hyderabaad
  - Nizam's Institute of Medical Sciences, Hyderabaad
  - Christian Medical College and Hospital, Ludhiana
  - Jaslok Hospital and Research Centre, Mumbai
  - KEM Hospital Research Centre, Pune
  - Kerala Institute of Medical Science, Trivandrum
- Poland (10):
  - Klinika Nefrologii Dzieciecej SPSK nr 1 ACK AMG, Gdansk
  - Katedra i Klinika Kardiologii Dzieciecej SK nr 6, Gornoslaskie Centrum Zdrowia Dziecka i Matki, Slaska AM, Katowice
  - II Katedra Pediatrii, Klinika Kardiologii Dzieciecej UM w Lodzi, Lodz
  - Klinika Nefrologii i Dializoterapii, Instytut Centrum Zdrowia Matki Polki, Lodz
  - Klinika Kardiologii i Nefrologii Dzieciecej AM, Poznan
  - I Klinika Chorob Dzieci SPSK nr 1 PAM, Szczecin
  - Oddzial Nefrologi Dzieciecej ze Stacja Dializ SSP ZOZ nad Dziecklem i Mlodzieza, Szczecin
  - Oddzial Pediatrii i Nefrologii ze Stacja Dializ, Wojewodzki Szpital Dzieciecy, Torun
  - Klinika Nefrologii i Transplantacji Nerek, Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw
  - Klinika Nefrologii Pediatrycznej AM, Wroclaw
- South Africa (9):
  - Benmed Park Clinic, Benoni
  - Chris Hani Baragwanath, Johannesburg
  - Global Clinical Trial Centre, Port Elizabeth
  - Potchefstroom Medi-Clinic, Potchefstroom
  - Eastmed Medical centre, Pretoria
  - Jubilee CTC Jubilee Hospital, Pretoria
  - Pretoria Academic Hospital, Pretoria
  - Zuid Afrikaans Hospital, Pretoria
  - Sandton Clinical Research Centre, Sandton
- Turkey (Türkiye) (4):
  - Istanbul University Istanbul Medical Faculty Pediatric Nephrology, Istanbul
  - Marmara University Medical Faculty Pediatric Nephrology, Istanbul
  - Dokuzeylul University Medical Faculty Pediatric Nephrology, Izmir
  - Ondokummayis University Medical Faculty Pediatric Nephrology, Samsun
- Ukraine (9):
  - Dnepropetrovsk Medical Academy, Department of Hospital Pediatrics on the bases of Regional Pediatric Hospital, Dnipro
  - Kharkov State University,Dept. of hospital pediatric on the bases of Regional Children's Hospital, Kharkiv
  - NMU n.b. Bogomolets, on b.o. Chil. Clin.Hosp.#2, Department of Pediatrics #2, Kiev
  - Institute of Pediatrics and Obstetrics AMS of Ukraine, Department of ecology related health problems, Kyiv
  - Danylo Halytskiy Lviv NationalMedical University, Department of Faculty, Lviv
  - Odessa State Medical University, Dept. of hospital pediatric and neonotology on the bases of Regional Children Hospital, Odesa
  - Crim.St. Med. Uni. On b.o. Rep. Child.Clin.Hosp. Chair of Pediat. W.c. of Physioth. Of the Postgr.dept, Simferopol
  - Uzhorod National University, Medical faculty, Department of Children's disease with course of Infection disease on the basis of City Children's Clinical Hospital., Uzhhorod
  - Vinnitsa National Medical Academy, Department of Hospital Pediatrics on the bases of Regional Pediatric Hospital, Vinnitsa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted from October 2006 to November 2007 at 56 international sites
Pre-assignment Details: Subjects entered placebo run-in prior to randomization
Period: Placebo Run-In
Arm/Group | Placebo | Ramipril Low Dose | Ramipril Mid Dose | Ramipril High Dose
Started | 422 | 0 | 0 | 0
Completed | 244 | 0 | 0 | 0
Not Completed | 178 | 0 | 0 | 0
Not completed — Did not meet blood pressure criteria | 119 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 19 | 0 | 0 | 0
Not completed — Reason not specified | 40 | 0 | 0 | 0
Period: Randomized
Arm/Group | Placebo | Ramipril Low Dose | Ramipril Mid Dose | Ramipril High Dose
Started | 83 | 41 | 40 | 80
Completed | 81 | 41 | 40 | 80
Not Completed | 2 | 0 | 0 | 0
Not completed — Did not receive study drug | 2 | 0 | 0 | 0
Period: Treated
Arm/Group | Placebo | Ramipril Low Dose | Ramipril Mid Dose | Ramipril High Dose
Started | 81 | 41 | 40 | 80
Completed | 79 | 40 | 40 | 76
Not Completed | 2 | 1 | 0 | 4
Not completed — Adverse Event | 1 | 0 | 0 | 2
Not completed — Reason not specified | 1 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ramipril Low Dose | Ramipril Mid Dose | Ramipril High Dose | Total
Number analyzed (Participants) | 81 | 41 | 40 | 80 | 242
Age Continuous [Mean (Standard Deviation); unit: years] | 12.2 (3.06) | 12.3 (3.03) | 12.1 (2.81) | 12.3 (3.06) | 12.2 (2.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 16 | 11 | 29 | 88
  Male | 49 | 25 | 29 | 51 | 154
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 21 | 11 | 10 | 20 | 62
  Asian | 8 | 1 | 4 | 10 | 23
  Caucasian | 27 | 15 | 13 | 29 | 84
  Hispanic | 25 | 14 | 13 | 20 | 72
  Other | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 4 Weeks in Trough Sitting Systolic Blood Pressure
Description: Value at end of treatment minus value at baseline, comparing the high-dose ramipril group with placebo
Time Frame: Baseline to 4 weeks
Population: Intent to treat (ITT) analysis including only treated participants who had at least one post-baseline assessment (1 placebo patient was treated but had no post-baseline assessment); last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Ramipril Low Dose | Ramipril Mid Dose | Ramipril High Dose
Number analyzed (Participants) | 80 | 41 | 40 | 80
mm Hg | -8.1 (7.92) | -9.7 (10.68) | -11.1 (8.88) | -11.3 (8.76)
Statistical Analysis 1: Comparison: Placebo vs Ramipril High Dose; Planned interim efficacy analysis: 80 placebo and 80 high-dose ramipril subjects provided 93% power, alpha=0.032, to detect 5 mmHg difference in primary outcome. SD of 8.5 mmHg assumed. Alpha of 0.032 required for the planned interim efficacy analysis. If study continued: 450 total subjects would provide 90% power, alpha=0.027, to detect 3 mmHg difference between placebo and combined ramipril dose groups. Alpha of 0.027 required for the final analysis; Test type: Superiority or Other; p = 0.044, ANCOVA — two-sided test; test from contrast statement from full model

2. Secondary Outcome: Change From Baseline to 4 Weeks in Trough Sitting Diastolic Blood Pressure
Description: Value at end of treatment minus value at baseline, comparing the high-dose ramipril group with placebo
Time Frame: Baseline to 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Ramipril Low Dose | Ramipril Mid Dose | Ramipril High Dose
Number analyzed (Participants) | 80 | 41 | 40 | 80
mm Hg | -5.0 (10.04) | -5.8 (10.17) | -6.1 (8.03) | -8.4 (9.14)
Statistical Analysis 1: Comparison: Placebo vs Ramipril High Dose; Test type: Superiority or Other; p = 0.006, ANCOVA — two-sided, unadjusted; test from contrast statement from full model

3. Secondary Outcome: Change From Baseline to 4 Weeks in Serum Creatinine
Description: Value at end of treatment (up to 4 weeks) minus value at baseline
Time Frame: Baseline up to 4 weeks
Population: Number of participants analyzed is less than number treated in the participant flow section because analysis includes only treated participants who had both a baseline and a post-baseline assessment; LOCF
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Ramipril Low Dose | Ramipril Mid Dose | Ramipril High Dose
Number analyzed (Participants) | 78 | 39 | 38 | 77
mg/dL | 0.04 (0.305) | 0.06 (0.275) | 0.03 (0.133) | 0.06 (0.211)

4. Secondary Outcome: Change From Baseline to 4 Weeks in Serum Potassium
Description: Value at end of treatment (up to 4 weeks) minus value at baseline
Time Frame: Baseline up to 4 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Ramipril Low Dose | Ramipril Mid Dose | Ramipril High Dose
Number analyzed (Participants) | 79 | 39 | 40 | 77
mg/dL | 0.01 (0.742) | -0.20 (0.475) | -0.08 (0.418) | 0.07 (0.559)

5. Secondary Outcome: Change From Baseline to 4 Weeks in Schwartz Formula Glomerular Filtration Rate (GFR)
Description: Value at end of treatment (up to 4 weeks) minus value at baseline; GFR is a measure of kidney function.
Time Frame: Baseline up to 4 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/min per 1.73 m2
Arm/Group | Placebo | Ramipril Low Dose | Ramipril Mid Dose | Ramipril High Dose
Number analyzed (Participants) | 78 | 39 | 38 | 77
mL/min per 1.73 m2 | -4.2 (27.85) | -6.0 (24.74) | -5.9 (26.29) | -6.9 (30.58)

ADVERSE EVENTS:
Arm/Group | Placebo | Ramipril Low Dose | Ramipril Mid Dose | Ramipril High Dose
Serious Adverse Events (participants affected / at risk) | 0/81 | 1/41 | 1/40 | 0/80
Other Adverse Events (participants affected / at risk) | 11/81 | 8/41 | 6/40 | 12/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | Ramipril Low Dose (N=41) | Ramipril Mid Dose (N=40) | Ramipril High Dose (N=80)
pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | Ramipril Low Dose (N=41) | Ramipril Mid Dose (N=40) | Ramipril High Dose (N=80)
abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 3 | 1
chest pain (General disorders) | 0 | 0 | 3 | 0
upper respiratory tract infection (Infections and infestations) | 2 | 4 | 1 | 1
dizziness (Nervous system disorders) | 2 | 0 | 2 | 2
headache (Nervous system disorders) | 6 | 4 | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agreed not to individually publish results of the study. Investigators may participate in a joint multicenter publication of the study results. Written notice must be provided to King. King has the right to review the publication and can require deletion of Confidential Information and delay of publication to allow for filing of patent applications.